CLINICAL TRIAL: NCT00990652
Title: A Phase II Trial Evaluating the Effects of Bortezomib in Patients With Recurrent Malignant Gliomas Treated Prior to Surgery and Then Bortezomib and Temozolomide Post-operatively
Brief Title: Presurgery Bortezomib for Recurrent Malignant Gliomas Followed by Postop Bortezomib & Temozolomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey Raizer, Jeffrey Raizer, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 08C5; STU00008280 (Other: Northwestern University IRB)
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Bortezomib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib + Temozolomide (Experimental): Patients receive an injection of bortezomib 1.7mg/m^2 on days 1, 4 and 8. Patients then undergo their standard of care surgery on day 8 or 9 to remove the tumor. Once recovered from surgery, patients receive combination treatment with temozolomide and bortezomib in periods called cycles (1 cycle = 28 days). Temozolomide is taken by mouth on days 1-7 and 14-21 of each cycle, and bortezomib injections are given on days 7 and 21 of each cycle.
  Interventions: Drug: Bortezomib; Drug: Temozolomide

INTERVENTIONS:
Drug: Bortezomib — Before surgery, an injection of bortezomib is given on days 1, 4, and 8. After surgery, bortezomib is given on days 7 and 21 of each cycle (1 cycle = 28 days).
  Other Names: Velcade
Drug: Temozolomide — After surgery, temozolomide is taken by mouth on days 1-7 and 14-21 of each cycle (1 cycle = 28 days).
  Other Names: Temodar

SUMMARY:
Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving bortezomib together with temozolomide after surgery may kill any tumor cells that remain after surgery.

This phase II trial is studying how well giving bortezomib before surgery followed by giving bortezomib together with temozolomide after surgery works in treating patients with recurrent malignant glioma.

DETAILED DESCRIPTION:
Patients receive bortezomib IV on days 1, 4, and 8. Patients then undergo surgical resection of the tumor on day 8 or 9.

Beginning approximately 14 days after surgery, patients receive oral temozolomide on days 1-7 and 14-21 and bortezomib IV on days 7 and 21. Treatment repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Tumor tissue and blood samples are collected periodically for biomarker analysis, gene methylation studies, and pharmacokinetic studies.

After completion of study therapy, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant glioma, including any of the following subtypes:

  * Glioblastoma multiforme
  * Gliosarcoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified
* Must show unequivocal evidence of tumor recurrence or progression by MRI or CT scan with contrast
* Candidate for surgery AND requires surgery

  * Evaluable or measurable disease following resection of recurrent tumor is not required
* Failed prior standard radiotherapy and temozolomide

  * Patients who have undergone stereotactic radiosurgery must have confirmation of true progressive disease (rather than radiation necrosis) by PET scan, magnetic resonance spectroscopy (MRS), or magnetic resonance perfusion (MRP) prior to surgery
  * Patients with lower-grade gliomas that have undergone radiographic malignant transformation allowed provided they failed radiotherapy (with or without temozolomide) and require surgery
* Life expectancy > 12 weeks

Exclusion Criteria:

* Not pregnant or nursing
* Negative pregnancy test
* No other medical issues (e.g., bleeding, infection, HIV, or serious medical or psychiatric illness) that would preclude study therapy
* Myocardial infarction within the past 6 months
* No other active cancer(s) except non-melanoma skin cancer or carcinoma in situ of the cervix, unless in complete remission and off of all therapy for that cancer for ≥ 3 years
* No hypersensitivity to bortezomib, boron, or mannitol
* More than 4 weeks since prior radiotherapy
* At least 4 weeks since prior cytotoxic therapy (6 weeks for nitrosoureas)
* At least 3 weeks since prior investigational drugs
* At least 2 weeks since prior enzyme-inducing anticonvulsants
* Concurrent non-enzyme-inducing anticonvulsants allowed
* No other concurrent standard or investigational anticancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Raizer, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened on May 21, 2009 with an accrual goal of 29 patients; the study was designed to enroll 10 patients initially and do an interim efficacy assessment. Accrual was suspended on February 11, 2011 for this analysis. The interim results did not support further accrual, and so the study was permanently closed to accrual on March 29, 2011.
Groups:
- Bortezomib + Temozolomide: Patients receive an injection of bortezomib 1.7mg/m^2 on days 1, 4 and 8. Patients then undergo their standard of care surgery on day 8 or 9 to remove the tumor. Once recovered from surgery (approximately 14 days later), patients receive combination treatment with temozolomide and bortezomib in periods called cycles (1 cycle = 4 weeks or 28 days). Temozolomide (75 mg/m^2) is taken by mouth on days 1-7 and 14-21 of each cycle, and bortezomib (1.3 mg/m^2) is given intravenously (IV) on days 7 and 21 of each cycle. Patients continue to receive cycles of treatment until disease progression, development of unacceptable toxicity, or up to a maximum of 24 months.
Period: Pre-surgical Bortezomib
Arm/Group | Bortezomib + Temozolomide
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1
Period: Surgical Resection
Arm/Group | Bortezomib + Temozolomide
Started | 9
Completed | 9
Not Completed | 0
Period: Post-sugery Bortezomib + Temozolomide
Arm/Group | Bortezomib + Temozolomide
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib + Temozolomide
Number analyzed (Participants) | 10
Age, Customized [Number; unit: participants]
  21-30 years | 0
  31-40 years | 0
  41-50 years | 6
  51-60 years | 2
  61-70 years | 2
  71-80 years | 0
  81-90 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Correlation of Expression of NFKBIA Gene With Response to Therapy and Survival.
Description: The effects of bortezomib on the endogenous modulators of NF-Kappa B pathways, especially the NFKBIA gene (nuclear factor of kappa light polypeptide gene enhancer in B-cells inhibitor, alpha) were assessed using novel assay technology; expression of NFKBIA was then correlated with response to therapy and patient survival.
Time Frame: Tissue samples for analysis were obtained on the day of surgery for all patients
Reporting Status: Not Posted

2. Primary Outcome: Number of Patients Surviving Without Disease Progression After 6 Months
Description: Patients will be monitored from date of first treatment to the date of first observation of progressive disease, non-reversible neurologic progression or increasing steroid requirements, death due to any cause, or early discontinuation of treatment. Progression-free survival will be defined as the absence of any of the above after 6 months.
  Progression (defined by MacDonald Criteria) is a 25% increase in the sum of products of all measurable lesions over smallest sum observed compared to baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to the cancer).
Time Frame: From date of first treatment until disease progression, death, or early discontinuation of treatment (up to 24 months)
Measure: Number; unit: participants
Arm/Group | Bortezomib + Temozolomide
Number analyzed (Participants) | 10
participants | 0

3. Secondary Outcome: Number of Participants Achieving a Response to Treatment (Either Complete or Partial Response) as Defined by MacDonald Criteria
Description: This measure was assessed only in patients who had residual tumor post-operatively. Per MacDonald Criteria:
  Complete Response requires complete disappearance of all measurable & evaluable disease, no new lesions, no evidence of non-evaluable disease, and only minimal or no use of steroids.
  Partial Response is defined as >= 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable lesions, no progression of evaluable disease, and no new lesions. Responders must be on the same or decreasing doses of steroid.
  Response was assessed by imaging (MRI or CT with contrast).
Time Frame: Day of treatment post-surgery and then approximately every 8 weeks thereafter until off treatment
Population: Only those participants who had residual tumor remaining after surgical resection were evaluated for this outcome.
Measure: Number; unit: participants
Arm/Group | Bortezomib + Temozolomide
Number analyzed (Participants) | 3
participants | 0

4. Secondary Outcome: Number of Grade 1, 2, 3, 4, and 5 Adverse Events Observed During Study Treatment (Defined by CTCAE v 3.0)
Description: Adverse events (AEs) were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0. In general, AEs are graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Days 1, 4, 8 pre-surgery, and then at the start of every cycle (approximately every 4 weeks) post-surgery while on treatment
Measure: Number; unit: adverse events
Arm/Group | Bortezomib + Temozolomide
Number analyzed (Participants) | 10
adverse events
  Grade 1 | 80
  Grade 2 | 30
  Grade 3 | 11
  Grade 4 | 1
  Grade 5 | 0

5. Other Pre Specified Outcome: Change in MGMT Methylation Status as Well as Other Methylation Patterns in Plasma
Description: To determine MGMT methylation status as well as other methylation patterns in plasma
Time Frame: Blood samples drawn on days 1, 4, and 8 pre-surgery, and then prior to cycle 1 and every 2 cycles thereafter
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Pharmacokinetics of Bortezomib in Tumor Tissue Taken at the Time of Surgery.
Time Frame: Tissue sample taken at the time of surgery for all patients.
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival (in Days)
Time Frame: Days 1, 4, 8 pre-surgery, once per cycle (every 4 weeks) while on treatment post-surgery, and then every 3 months up to 2 years during follow-up
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bortezomib + Temozolomide
Number analyzed (Participants) | 10
days | 248 [122 to 397]

8. Secondary Outcome: Overall Survival Rate at 6 Months
Description: The rate of overall survival at 6 months (regardless of disease progression) was calculated.
Time Frame: After 6 months on study
Population: The 6-month overall survival rate was based on a median of 168 days of follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib + Temozolomide
Number analyzed (Participants) | 10
percentage of participants | 69

ADVERSE EVENTS:
Description: Adverse events were assessed by exam, lab tests, and review with patients during study visits.
Arm/Group | Bortezomib + Temozolomide
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Bortezomib + Temozolomide (N=10)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hemorrhage, CNS (Nervous system disorders) | 1 (1)
Infection with normal ANC (Infections and infestations) | 1/7 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib + Temozolomide (N=10)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (6)
Leukocytes decreased (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4)
Platelets (Blood and lymphatic system disorders) | 5 (5)
Cardiac General - Other (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
INR elevated (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (6)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis -oral cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Infection with unknown ANC - wound (Infections and infestations) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1)
ALT, SGPT elevated (Metabolism and nutrition disorders) | 6 (6)
AST, SGOT elevated (Metabolism and nutrition disorders) | 4 (4)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (4)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (6)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 3 (3)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Memory impairment (Nervous system disorders) | 1 (1)
Mood alteration - Anxiety (Nervous system disorders) | 1 (1)
Mood alteration - Depression (Nervous system disorders) | 2 (2)
Neuropathy: cranial - CN II Vision (Nervous system disorders) | 1 (1)
Neuropathy: cranial - CN VII Motor-face; Sensory-taste (Nervous system disorders) | 1 (1)
Neuropathy: cranial - CN XI Motor-sternomastoid and trapezius (Nervous system disorders) | 1 (1)
Vision-blurred vision (Ear and labyrinth disorders) | 1 (1)
Pain - Head/headache (General disorders) | 5 (5)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes